CLINICAL TRIAL: NCT00164775
Title: The Efficacy of Imipramine in Treatment of Functional Dyspepsia: A Double Blind Randomized Placebo Controlled Trial
Brief Title: The Efficacy of Imipramine in Treatment of Refractory Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Justin Che-Yuen Wu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA Study
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Functional Gastrointestinal Disorder
Keywords: Functional dyspepsia, refractory, antidepressant
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Imipramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imipramine (Active Comparator): Imipramine 25mg nocte for first 2 weeks then Imipramine 50 mg nocte for 10 weeks
  Interventions: Drug: Imipramine
- Placebo (Placebo Comparator): Placebo 1 tablet for first 2 weeks then Placebo 2 tablets for 10 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imipramine — 25mg nocte for first 2 weeks then 50 mg nocte for 10 weeks
  Arms: Imipramine
Drug: Placebo — One tab nocte for first 2 weeks then 2 tabs for 10 weeks
  Arms: Placebo

SUMMARY:
The aim of this study is evaluate the efficacy of Imipramine, a tricyclic antidepressant, in treatment of functional dyspepsia. This is a double blind randomised placebo controlled trial in which consecutive patients with diagnosis of functional dyspepsia will be studied. After exclusion of organic cause of dyspepsia by endoscopy, these patients will be randomly assigned to either imipramine or placebo. All the patients will enter an additional 4 weeks of drug withdrawal phase after the initial 12 weeks of study drug treatment. They will be evaluated for treatment response, which is defined as satisfactory relief of dyspeptic symptoms at the end of 12-week treatment.

DETAILED DESCRIPTION:
Functional dyspepsia is a heterogeneous disorder that consists of a variety of upper gastrointestinal symptoms such as postprandial fullness, early satiety, pain, bloating, belching, or nausea. The pathophysiology of functional dyspepsia is not fully understood and the correlation of those proposed mechanisms with the clinical characteristics and treatment response is poor. Owing to the poor understanding on the mechanism, treatment of functional dyspepsia has been far from satisfactory. There are numerous modalities of medical treatment that has been reported to be effective but the results are conflicting. Large and well-controlled studies in functional dyspepsia have shown that proton pump inhibitor had a therapeutic gain of about 10%-15% better than placebo in patients with functional dyspepsia. However, this positive effect was restricted to patients with reflux-like dyspepsia, a subgroup that actually is no longer considered to belong to functional dyspepsia. Prokinetic agent is another class of drug that has been widely used in functional dyspepsia. Although recent reviews suggest that prokinetics are more effective than placebo, most trials were flawed with significant heterogeneity among studies. Tricyclic antidepressant (TCA) is another important class of drug that is commonly used in various functional gastrointestinal disorders (FGID) and chronic pain disorders. The effectiveness of TCA in FGID has been supported by a meta-analysis, which reported that improvement in global GI symptoms against placebo was highly significant. The mechanism of TCA in treatment of FGID is poorly understood but the therapeutic effect is evident even in low dose, suggesting that it is independent of its anti-depressive action. To date, clinical trial of TCA in treatment of FD with sufficient sample size and well-defined clinical endpoint is still lacking. So the objective of this study is to evaluate the efficacy of imipramine, a tricyclic antidepressant, in treatment of functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfill the diagnostic criteria of functional dyspepsia as defined by Rome II criteria
* Age > 18 years old
* Failure of treatment response to PPI, H2 receptor antagonist fo 8 weeks and domperidone for 4 weeks

Exclusion Criteria:

* Organic pathology detected by endoscopy
* GERD or IBS as dominant compliant
* Presence of any alarm symptom: anemia, recurrent vomiting, weight loss
* Concomitant Helicobacter pylori infection
* Concomitant use of neuroleptic or antidepressant, NSAID
* Previous gastrointestinal surgery
* Cardiac arrhythmia, untreated glaucoma or benign prostate hypertrophy
* Pregnancy
* Known hypersensitivity or contraindication for tricyclic antidepressant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2005-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Overall satisfactory relief (Global Symptom Assessment) at 12 weeks | 12 weeks
  It is defined as a response of "Yes" to the question: "Do you experience overall satisfactory relief of dyspeptic symptom with the current treatment?" by global symptom assessment.

SECONDARY OUTCOMES:
Individual dyspeptic symptom scores | 12 weeks
  8-item dyspepsia symptom score questionnaire assessing epigastric pain, epigastric burning, postprandial fullness, early satiety, belching, bloating, nausea, and vomiting on a scale of 0-3 over the last 7 days
Days of sleep disturbance | 12 weeks
  Effect on sleep will be assessed by asking patients if they had insomnia on ≥1 day per week
Mood assessment | 12 weeks
  Effect on mood will be assessed using the hospital anxiety and depression scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Justin CY Wu, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheong PK, Ford AC, Cheung CKY, Ching JYL, Chan Y, Sung JJY, Chan FKL, Wu JCY. Low-dose imipramine for refractory functional dyspepsia: a randomised, double-blind, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2018 Dec;3(12):837-844. doi: 10.1016/S2468-1253(18)30303-0. Epub 2018 Oct 22. PMID 30361080